# National

# **Cardiogenic Shock Initiative**

Version 3.0 July, 2018





# National Cardiogenic Shock Initiative (NCSI, National CSI)

# **STUDY SPONSOR:**



# **Henry Ford Health System**

2799 W. Grand Blvd.
Center for Structural Heart Disease - CFP # 439
Detroit, Michigan 48202
(313) 916-8708
NationalCSI@hfhs.org

# **PRINCIPLE INVESTIGATOR:**

William W. O'Neill, MD, FACC, FSCAI

Henry Ford Health System 2799 W. Grand Blvd. Center for Structural Heart Disease - CFP # 439 Detroit, Michigan 48202 (313) 916-8708

# **TABLE OF CONTENTS**

| | | Page |
|---|---|---|
| • | Introduction | 4 |
| • | Research Procedures | 6 |
| • | Quality Metrics | 6 |
| • | Population and Eligibility | 7 |
| • | Risks/Benefits/Alternatives | 8 |
| • | Data Management | 9 |
| • | Access to Patient Information | 10 |
| • | Analysis and Publication of Data | 10 |
| • | Appendix 1: NSCI Treatment Algorithm (Standard Care) | 12 |
| • | Appendix 2: Adoption of the NCSI Treatment Algorithm & Joining the NCSI | 16 |
| • | Appendix 3: Case Report Form (CRF) | 18 |
| • | Appendix 4: Patient Exclusion Form (PEF) | 24 |
| • | Appendix 5: 30 Day Month Follow-up Form | 26 |
| • | Appendix 6: 1 Year Follow-up Form | 27 |

# Introduction

Acute myocardial infarction complicated by cardiogenic shock (AMICS) is a deadly condition with a historical in-hospital survival of only 50%<sup>1-3</sup>. To date, the only therapy proven to benefit patients in AMICS using data from randomized control trials has been early mechanical reperfusion<sup>3</sup>. Accordingly, current American and European guidelines confer a class IB indication for reperfusion therapy in the setting of AMICS<sup>4</sup>. Unfortunately, little progress has been made on improving survival with subsequent therapies, including intra-aortic balloon pump counter-pulsation (IABP) <sup>5</sup>. This lack of progress is worrisome since the incidence of AMICS appears to be increasing<sup>6-7</sup>.

With the FDA approval of Impella (Abiomed, Danvers, MA) in AMICS, a powerful new tool has become available for hemodynamic support. Impella is a transcatheter axial flow pump, delivered percutaneous, with the ability to provide 2.5 to 4.0 liters/minute of forward flow. The device should provide sufficient forward cardiac flow to support vital organs in the majority of patients who present with AMICS. Since Impella is the only percutaneous temporary ventricular support device approved as safe and effective for use in AMICS, the use of the device has steadily grown<sup>8</sup>. Unfortunately, there is little data available to providers as to the best practice patterns associated with the delivery and use of Impella in AMICS. In fact, a retrospective analysis of 15,259 patients treated with an Impella between 2009 and 2017 revealed a wide variety of outcomes associated with the use of Impella in AMICS, with approximately one third of hospitals having a survival rate of 25%, another third of hospitals having a survival rate of 50%, and yet another third of hospitals having a survival rate of 75%.

In the summer of 2016, cardiologists from four highly competitive healthcare systems in southeast Michigan came together in an attempt to increase survival in patients who present with

AMICS. Leaders from each healthcare system debated and discussed key elements in the improvement of care for patients who present with AMICS. Using the most up-to-date research, a treatment algorithm for AMICS was developed and subsequently implemented as a quality improvement initiative throughout southeast Michigan. Patient information was gathered by each of the sites and collected in a retrospective registry. Outcomes and results were shared during quarterly meetings and concluded with a 41-patient pilot feasibility study. This initial pilot study revealed a 76% survival to discharge, a significant improvement compared to prior historical controls.

Given the promising outcomes, leaders from around the world have implemented the treatment algorithm in their local clinical practices with similar results. We have therefore launched the National Cardiogenic Shock Initiative (NCSI). The aim of the NCSI is to bring together experienced centers across the nation who are experts in mechanical reperfusion therapies and have a large experience with the use of mechanical circulatory support devices to systematize care in AMICS. Our goal is to dramatically decrease the duration patients remain in cardiogenic shock and attempt to decrease total usage and duration of vasopressors and ionotropic agents. We aim to further demonstrate that rapid delivery of mechanical circulatory support will improve hemodynamics, reverse the spiraling neuro-hormonal cascade associated with cardiogenic shock, allowing clinicians to decrease use of vasopressors and inotropic agents and ultimately improve survival.

Healthcare systems that have agreed to adopt the NCSI treatment algorithm are being asked to participate in this prospective registry so that patient outcomes can be analyzed (see Appendix 2). Participating investigators will be asked to voluntarily provide data from patients completing the treatment algorithm to be included in the NCSI Registry.

# **Research Procedures**

After a patient has been treated according to the NCSI treatment algorithm at the discretion of their physician (see Appendix 1), they will be approached prior to discharge and asked to participate in NCSI registry, including obtaining permission to allowing coordinators to conduct a 1-month and 1-year follow-up. This data collection can occur via follow up phone call, electronic chart review, or any other method that complies with the site's SOPs. If the patient is discharged prior to obtaining consent, consent form and explanation of the study can be mailed to the patient for their signature and return. If more than one (1) year has passed, all data may be obtained retrospectively.

If consent is provided, then the following data will be collected (see case report form - Appendix 3):

# **Retrospective Data (from their medical records)**

- Medical history
- Admission characteristics
- Procedure dates and times
- Procedure characteristics
- Diagnostic values
- Post-procedure information

# **Prospective Data (from follow-up)** (see Appendix 5 and Appendix 6)

- Mortality at 1 month from AMICS
- Mortality at 12 months from AMICS

From this data, the following Quality Metrics will be tracked:

- Discharge survival
- Duration of shock-to-support times

- Use of Impella Support pre-PCI
- Use of right heart catheter for hemodynamic monitoring
- Attainment of TIMI III flow post reperfusion
- Attainment of Cardiac power > 0.6 watts after completion of therapy
- Reduction or elimination of vasopressors and inotropic agents.

# Population and Eligibility Criteria

Due to the heterogeneous cohort of patients who present with AMICS, we have defined a specific subset of patients from whom outcomes are to be collected. Approximately 500 adult patients will be approached to participate in the registry at approximately 75 sites in the United States. The duration of hospital participation in this research study is anticipated to be approximately 3 years.

# **Registry Inclusion Criteria**

- Symptoms of acute myocardial infarction (AMI) with ECG and/or biomarker evidence of S-T elevation myocardial infarction (STEMI) or non-S-T elevation myocardial infarction (NSTEMI)
- 2. Cardiogenic shock is defined as the presence of at least two of the following:
  - a. Hypotension (systolic blood pressure ≤90 mm Hg, or inotropes/vasopressors to maintain systolic blood pressure ≥90 mmHg)
  - b. Signs of end organ hypoperfusion (cool extremities, oliguria or anuria, or elevated lactate levels)
  - c. Hemodynamic criteria represented by a cardiac index of <2.2 L/min/m² or a cardiac power output ≤0.6 watts.

- 3. Patient is supported with an Impella
- 4. Patient undergoes PCI

# **Registry Exclusion Criteria**

- 1. Evidence of Anoxic Brain Injury
- 2. Unwitnessed out of hospital cardiac arrest or any cardiac arrest in which return of spontaneous circulation (ROSC) is not achieved within 30 minutes
- 3. IABP placed prior to Impella
- 4. Septic, anaphylactic, hemorrhagic, and neurologic causes of shock
- 5. Non-ischemic causes of shock/hypotension (pulmonary embolism, pneumothorax, myocarditis, tamponade, etc.)
- 6. Active bleeding for which mechanical circulatory support is contraindicated
- 7. Recent major surgery for which mechanical circulatory support is contraindicated
- 8. Mechanical complications of AMI (acute ventricular septal defect (VSD) or acute papillary muscle rupture)
- Known left ventricular thrombus for which mechanical circulatory support is contraindicated
- 10. Mechanical aortic prosthetic valve
- 11. Contraindication to intravenous systemic anticoagulation

# Risks/Benefits of and Alternatives to Patient Participation

This is not a treatment study. This is a single-arm prospective registry that captures data generated during procedures which are considered standard of care using FDA-approved technology. There are no risks other than breach of confidentiality. To mitigate this risk, patient identifiers are not being captured, and all data will be stored in a secure REDCap database

(please see below). There are no benefits in participation other than the scientific knowledge gained, and the only alternative to participation is not participating.

# **Data Management**

Data collected by the participating sites will be stored and managed in a secure REDCap study database hosted through the Henry Ford Health System Department of Public Health Sciences in Detroit, Michigan. REDCap (Research Electronic Data Capture) is a secure, webbased application designed to support data capture for research studies. A specific database was created solely for NCSI in September 2017. The REDCap database that was custom-built for this study includes only the specific data fields that pertain to the data points being collected in the study, which are present on the case report form (CRF) (see Appendix 3).

For patients who present to affiliated hospitals with AMICGS but are excluded from entry into the registry, a Patient Exclusion Form will be sent to track the reasons for exclusion (see Appendix 4).

The CRFs and Patient Exclusion Forms from an individual site will be transmitted to the lead site, Henry Ford Hospital, via secure email and accessed only on hospital-approved, password-protected computers and stored on a password-protected and encrypted OneDrive system by Microsoft. Access to the OneDrive system and the REDCap database will be managed at the lead site by the NCSI coordinator and the investigators of the study via hospital-approved, password-protected computers inside locked offices in Henry Ford Hospital.

# **Access to Patient Information**

The following will have access to the de-identified patient medical information, and any necessary research contracts and Data Use Agreements will be completed for each participating site.

Henry Ford Hospital – Detroit, Michigan:

- The NCSI team:
  - o PI
  - Co-Investigator
  - NCSI Coordinator
  - Research Nurse
  - Research Assistant
  - Data Coordinator
- Statistician, based at Henry Ford Hospital

# **Analysis and Publication of Data**

There will be planned interim analysis of the data for the purpose of presentation as well as a final analysis and submission for publication of all data at the end of the study enrollment and follow-up.

# References

- 1. Goldberg, R. J., Makam, R. C. P., Yarzebski, J., McManus, D. D., Lessard, D., & Gore, J. M. (2016). Decade-Long Trends (2001–2011) in the Incidence and Hospital Death Rates Associated with the In-Hospital Development of Cardiogenic Shock after Acute Myocardial Infarction. *Circulation: Cardiovascular Quality and Outcomes*, 9(2), 117-125.
- 2. Kolte D, Khera S, Aronow WS, Mujib M, Palaniswamy C, Sule S, Jain D, Gotsis W, Ahmed A, Frishman WH, Fonarow GC. Trends in incidence, management, and outcomes of cardiogenic shock complicating ST-elevation myocardial infarction in the United States. J Am Heart Assoc. 2014 Jan 13;3(1):e000590
- 3. Hochman, J. S., Sleeper, L. A., White, H. D., Dzavik, V., Wong, S. C., Menon, V., & Boland, J. (2001). One-year survival following early revascularization for cardiogenic shock. *JAMA*, 285(2), 190-192.
- 4. Bainey, K. R., & Armstrong, P. W. (2016). Transatlantic Comparison of ST-Segment Elevation Myocardial Infarction Guidelines: Insights From the United States and Europe. *Journal of the American College of Cardiology*, 67(2), 216-229.
- 5. Thiele H., Zeymer U., Neumann F.J., et al.(2012) Intraaortic balloon support for myocardial infarction with cardiogenic shock. N Engl J Med 367:1287–1296
- 6. Center for Medicare and Medicaid database, MEDPAR FY14
- 7. Killip, T., & Kimball, J. T. (1967). Treatment of myocardial infarction in a coronary care unit: a two year experience with 250 patients. *The American journal of cardiology*, 20(4), 457-464.
- 8. Stretch R, Sauer C.M., Yuh D.D., Bonde P.(2014) National trends in the utilization of short-term mechanical circulatory support: incidence, outcomes, and cost analysis. J Am Coll Cardiol 64:1407–1415.
- William O'Neill, Mir Basir, Simon Dixon, Kirit Patel, Theodore Schreiber, Steven Almany. Feasibility of Early Mechanical Support During Mechanical Reperfusion of Acute Myocardial Infarct Cardiogenic Shock JACC: Cardiovascular Interventions Mar 2017, 10 (6) 624-625

# **NSCI Treatment Algorithm**

### 1. Confirmation of AMI Shock

The diagnosis of AMI is confirmed by electrocardiographic changes indicative of new or presumed new ischemia (new ST-T wave changes), detection of elevated cardiac biomarkers or angiographic findings of an infarct related artery on coronary angiogram in the presence of ischemic symptoms.

Cardiogenic shock is defined as the presence of at least two of the following:

- Hypotension (systolic blood pressure ≤90 mm Hg, or inotropes/vasopressors to maintain systolic blood pressure ≥90 mmHg)
- 2. Signs of end organ hypoperfusion (cool extremities, oliguria or anuria, or elevated lactate levels)
- 3. Hemodynamic criteria represented by a cardiac index of <2.2 L/min/m<sup>2</sup> or a cardiac power output  $\le$ 0.6 watts.

# 2. Access, Baseline Invasive Hemodynamics

Due to the heterogeneous cohort of patients who present with AMICS, any diagnostic steps to ensure the presence of AMI or CS are left to the discretion of the primary operator (ie: timing of right heart catheterization, coronary angiogram and placement of MCS). We do recommend obtaining femoral access to ensure adequate vessel size for MCS. If a right heart catheterization has not been performed prior to MCS placement we recommend measuring a LVEDP prior to placement of MCS. In the event a LVEDP ≤15 mmHg, an alternate diagnosis should be suspected and right heart catheterization should be performed prior to MCS to confirm presence of cardiogenic shock. Following placement of large-bore access and administration of systemic anticoagulation an Impella catheter will be inserted and manipulated to obtain maximum

forward flow. Right heart catheterization (RHC) will be performed for calculation of cardiac power output (CPO), SVR and PCWP/RA ratio and pulmonary artery pulsatility index (PAPi), during the index procedure.

# 3. Intervention

PCI of the culprit lesion(s) should be performed, per national recommendations. We recommend against non-culprit PCI unless flow is impaired in the involved artery (ie. less than TIMI 3 flow and excluding chronic total occlusions); however the ultimate decision of multivessel PCI lies with primary operator. PCI can be performed with thrombectomy if a heavy thrombus burden is present. Once appropriately sized stents have been implanted angiography will be performed to assess TIMI flow. If TIMI III flow is not present, intracoronary vasodilatory should be administered at the discretion of the primary operator.

Prior to discharge from the cath lab, a formal neurovascular check should be performed for assessment of Impella-related limb ischemia. This can be performed either by an in-depth physical examination, peripheral angiogram, or lower extremities doppler studies. If signs of limb ischemia are noted, the peel-away sheath should be removed (if not already done so) with reassessment. If limb ischemia persists, antegrade access should be performed to provide distal lower extremity blood flow.

# 4. Post-PCI Hemodynamics

After the intervention is completed, right heart pressures, cardiac output, and CPO will be obtained. If CPO is > 0.6, no further intervention is required. If CPO is  $\leq 0.6$ , right heart pressure will be reviewed to identify evidence of right ventricular failure if present (PAPi < 0.9).

If evidence of right ventricular failure are present (PAPi < 0.9), or if the Impella is suctioning, operators should consider right ventricular support with commercially available devices (Impella or Tandem Heart). Irrespective of CPO, evidence of RV shock is a warning not NCSI-Protocol-(v3.0)-July, 2018

to increase alpha agonists. These agents dramatically increase pulmonary vascular resistance (PVR) at a time of minimal RV reserve and can cause a lethal spiral as increasing doses of alpha agonists to maintain arterial pressure leads to decrease forward RV flow and worsens hypotension.

If CPO < 0.6 persists and RV shock is not the cause, consideration for the placement of an Impella 5.0 or a durable left ventricular assist device (LVAD) should be considered.

# 5. Weaning and Explantation

Impella devices should only be considered for explantation once the following criteria have been met:

- 1. Weaning of all inotropes and vasopressors
- 2. CPO > 0.6 watts without vasopressors or inotropes, and
- 3. PAPi > 0.9.

# 6. Safety and Monitoring

Cautious attention should be paid to the infrequent yet serious complication of limb ischemia with the use of large bore sheaths and devices. Detailed neurovascular checks should be performed while on Impella support. Use of antegrade sheaths to provide flow to the affected limb is strongly recommended in such cases. Prophylactic use antegrade access may also be considered, especially in patients who will likely require >24 hours of support. Although rare hemolysis can also occur, daily hemoglobin level should be obtained while on support. If there are signs of hematuria, Impella positioning should be checked via echocardiography.

# NATIONAL CARDIOGENIC SHOCK INITIATIVE ALGORITHM INCLUSION CRITERIA Acute Myocardial Infarction: STEMI or NSTEMI EKG and/or biomarker evidence of AMI (STEMI or NSTEMI) varies 3400K potension (<90/60) or the need for vasopressors or inotropes to maintain systolic and pressure >90

# **EXCLUSION CRITERIA**

- Evidence of Anoxic Brain Injury
  Unwitnessed out of hospital cardiac arrest or any cardiac arrest in which ROSC is not achieved in 30 minutes
- IABP placed prior to Impella
- Septic, anaphylactic, hemorrhagic, and neurologic causes of shock Non-ischemic causes of shock/hypotension (Pulmonary Embolism, Pneumothorax, Myocarditis, Tamponade, etc.)

- Recent major surgery
  Mechanical Complications of AMI
  Known left ventricular thrombus
  Patient who did not receive revascularization
- Contraindication to intravenous systemic anticoagulation
- Contraindication
   Mechanical aortic valve

# ACTIVATE CATH LAB

Evidence of end organ hypoperfusion (cool extremities, oliguria, lactic acidosis)

### ACCESS & HEMODYNAMIC SUPPORT

- Obtain femoral arterial access (via direct visualization with use of ultrasound and fluoro)
- Obtain venous access (Femoral or Internal Jugular) Obtain either Fick calculated cardiac index or LVEDP

IF LVEDP > 15 or Cardiac Index < 2.2 AND anatomy suitable, place IMPELLA

# \*\* QUALITY MEASURES \*\*

- Impella Pre-PCI
- Door to Support Time < 90 minutes
- Establish TIMI III Flow
- Right Heart Cath
- Wean off Vasopressors & Inotropes
- Maintain CPO > 0.6 Watts
- Improve survival to discharge to >80%

## Coronary Angiography & PCI

- Attempt to provide TIMI III flow in all major epicardial vessels other than CTO
- If unable to obtain TIMI III flow, consider administration of intra-coronary

# Perform Post-PCI Hemodynamic Calculations 1. Cardiac Power Output (CPO): MAP x CO

2. Pulmonary Artery Pulsatility Index (PAPI): sPAP - dPAP

### Wean OFF Vasopressors and Inotropes

If CPO is >0.6 and PAPI >0.9, operators should wean vasopressors and inotropes and determine if Impella can be weaned and removed in the Cath Lab or left in place with transfer to ICU.

### **Escalation of Support**

If CPO remains <0.6 operators should consider the following options:

PAPI is <0.9 consider right sided hemodynamic support

- PAPI >0.9 consideration for additional hemodynamic support Local practice patterns should dictate the next steps:
  - Placement of more robust MCS device(s) Transfer to LVAD/Transplant center
- If CPO is >0.6 and PAPI <0.9 consider providing right sided hemodynamic support if clinical suspicion for RV dysfunction/failure

### Vascular Assessment

- Prior to discharge from the Cath Lab, a detailed vascular exam should be performed including femoral angiogram and Doppler assessment of the affected limb.
  - If indicated, external bypass should be performed.

- ICU Care Daily hemodynamic assessments should be performed, including detailed vascular
- Monitor for signs of hemolysis and adjust Impella position as indicated

Device Weaning Impella should only be considered for explantation once the following criteria are met:

- Weaning off from all inotropes and vasopressors
- CPO > 0.6, and PAPI > 0.9

### Bridge to Decision

Patients who do not regain myocardial recovery within 3-5 days, as clinically indicated, should be transferred to an LVAD/Transplant center. If patients are not candidates, palliative care options should be considered.

# NATIONAL CARDIOGENIC SHOCK INITIATIVE

NationalCSI@hfhs.org

www.henryford.com/cardiogenicshock

NationalCSI - Algorithm - v1.5 - 11/2017

# Adoption of the NCSI Treatment Algorithm & Joining the NCSI

Adoption to the NCSI treatment algorithm is completely voluntary. Deviation from the treatment algorithm can occur without consultation of the primary investigators at the discretion of the primary operator. All AMICS patients, including those with treatment algorithm deviation, can be included in the NCSI registry as there is no formal, nationally accepted or standardized protocol or treatment algorithm for treatment of AMICS. Operators and hospitals are encouraged to review the pilot study data and treatment algorithm to determine if they wish to adopt the NCSI treatment algorithm as their standard of care for the treatment of AMICS.

Multi-hospital collaboration is considered a cornerstone to the success of the NCSI. We are reaching out nationally and encouraging hospitals to work together to collect data and demonstrate the success of regional shock protocols and/or treatment algorithms. Hospitals joining the NCSI group voluntarily agree to share data, post-discharge, including demographics, procedural characteristics and outcomes as detailed in the case report form. Data is de-identified and HIPAA-compliant. Data generated from the index procedure admission to discharge (or death, if prior to discharge) will be collected retrospectively and de-identified. Prior to discharge, surviving patients will be asked to consent to the collection of data at 30 days and 1 year post-index procedure. This data collection can occur via follow up phone call, electronic chart review, or any other method that complies with the site's SOPs.

To formally join and affiliate with NCSI, we request the minimum following requirements of the interested hospitals:

1. Implantation of >10 Impella per year (for any indication)

- 2. Adoption of the NCSI treatment algorithm as standard of care for patients who present with AMICS
- 3. Identification of a local Primary Investigator (PI) to coordinate data collection

  After the above requirements are met, a hospital may request to join NCSI through Henry Ford

  Hospital's NCSI website (www.henryford.com/cardiogenicshock). The hospital site will be

  contacted and interviewed by a member of the NCSI team. Once a hospital is accepted to join

  NCSI, a formal data-use agreement between the institution and Henry Ford Hospital must be

  completed.

# **Case Report Form**

# National Cardiogenic Shock Initiative Case Report Form

(Version 2.0)

Please complete the entirety of the worksheet. Upon completion, please email this worksheet [SECURE] to: NationalCSI@hfhs.org. Please email/call if there are any questions or concerns. Demographics Date of Impella Insertion Implanting Physician Hospital: Name Hospital: City, State Age of Patient Gender (please circle) Female Male Race (please circle) White Black Hispanic Other Medical History Does the patient have a history of Diabetes? Yes No N/A Doe the patient have a history of TIA/CVA? Yes No N/A Does the patient have a history of ESRD? Yes No N/A Does the patient have a history of CKD? Yes No N/A Does the patient have a known LVEF <50%? Yes No N/A Has the patient had a prior CABG? Yes No N/A Has the patient had a prior PCI? Yes No N/A Has the patient had a prior Myocardial Infarction? Yes No N/A

| FOR HFH USE ONLY |
|------------------|
| NCSI #: |

| Was the patient transferred from anothe | | Yes | No | N/A |
|---|---|---|---|---|
| If yes, was the patient on support<br>prior to transport? | | Yes | No | N/A |
| What support device was used? | | IABP | Other: | |
| Was cardiogenic shock present on admiss | sion | | | |
| to your institution? | | Yes | No | N/A |
| Did the patient experience any of the | | | | |
| following (prior to arrival in the Cath Lab)<br>Anoxic Brain Injury? | ): | Yes | No | N/A |
| Cardiac Arrest (In Hospital)? | | Yes | No | N/A |
| Cardiac Arrest (Out of Hospital)? | | Yes | No | N/A |
| Did the patient require CPR prior to Impe | ella implant? | Yes | No | N/A |
| Was the patient undergoing active CPR | | | | |
| at the time of Impella implantation? | | Yes | No | N/A |
| Was the patient treated with medically-in | nduced | V | No | N1/A |
| hypothermia? | | Yes | INO | N/A |
| ** Important Timings ** Please estin | nate if exact tir | nings are un | available. | |
| Please | do not leave b | olank. | | |
| Arrival to Hospital (date and time) | Date | 1 | Time | |
| Onset of AMI (date and time) | Date | 1 | Time | |
| Onset of Shock (date and time) | Date | 1 | Time | |
| Time of Impella Insertion (date and time) | Date | 1 | Time | |
| | the following t | rimes: | | |
| Using the above timings, please calculate | | | _ | |
| Using the above timings, please calculate Door to Support Time (minutes): | | | | |

2

National CSI – Case Report Form – (v2.0) – July, 2018

| RHC Placement: | nt: 1. Prior | to PCI | Post PCI 3. Intra-procedural | | | | |
|---|---|---|---|---|---|---|---|
| | 1. Prior | to Impella | 2. Post Impell | la | 3. No | RHC obtained | |
| Impe | lla Used: | Impella | Access: | | | AMI Type? | |
| 2.5 CP | 5.0 RP | | | | | | |
| Other: | | ☐ Femoral ☐ Other: | □Axillary | | | STEMI NSTEMI | |
| PCI Attempted? | TIMI FLOW | Evidence of | # of Diseased | # Vessels | # of | Culprit Lesion(s) | Other Lesion(s) |
| YES | D DOL D . DOL | Thrombus | Vessels? | Treated? | Stents? | Location(s) | Location(s) |
| NO | Pre-PCI Post-PCI | Pre-PCI? | | _ | | 1. LM 5. Ramus | 1. LM 5. Ramus |
| Successful? | 0 0 | YES | 0<br>1 | 0<br>1 | | 2.LAD 6. SVG | 2.LAD 6. SVG |
| YES | 2 2 | 123 | 2 | 2 | | 3. LCx 7. LIMA | 3. LCx 7. LIMA |
| NO | 3 3 | NO | 3 | 3 | | 4. RCA 8. RIMA | 4. RCA 8. RIMA |
| Access for PCI? | Was complete | Thrombectomy | Atherectomy | PCI Compli | cations? | □ NO □YES | |
| | revascularization | used? | used? | r Ci Compii | If YES: | Stent Thron | nbosis |
| 1. Radial | performed? | | | | | | Residual Thrombus |
| ļ | | | | | | □ OTHER: | |
| 2. Femoral | YES NO | YES NO | YES NO | | | | |
| Was patient takin | ng antiplatelet medica | ation at home? $\square$ | - | | el 🗆 Ticago | relor 🗆 Prasugrel 🗆 I | N/A |
| | | _ | OTHER:_ | | | | |
| Was patient load | ed with antiplatelet p | | | | _ | | , |
| | | □ Eftit | ibatide 🗆 Tirofil | ban □ N/A | ☐ OTHER: | | |
| f oral antiplatele | ts were given, what r | oute were they giv | /en? ☐ By Mout | h □ NG/OG | Tube 🗆 R | ectal N/A Othe | er: |
| Was the oral anti | platelet crushed? | Yes □ No □ N/A | | | | | |
| When was antiple | atelet administered? | □ EMS □ ER □ | Pre-PCI ☐ Post- | PCI ∐ N/A | ⊔ Other: _ | | |
| Anticoagulation u | used during PCI: 🗆 H | eparin 🗆 Bivaliru | din 🗆 Other: | | | | |
| Pleas | e give a brief desc | ription of the p | atient admiss | ion: | | | |

| HEMODYNAMIC & LAB | ORATORY VALUES (Pre-p | rocedure & Prior to starti | ng Vasoactive Medications) |
|---|---|---|---|
| These values should rep | present the "worst hemo | dynamics" that demonstra | te level of shock |
| HR | SBP | DBP | MAP |

| | | | dynamics prior | | | | | |
|---|---|---|---|---|---|---|---|---|
| HR | SBP | DBP | MAP | Troponin | Cr | AST | Hgb | Lactate |
| RA/CVP | RV | PA | PCWP | co | CI | CPO | PAPI | LVEDP |
| | | | | ☐ Fick ☐ TD | | | | |
| | | | | □ cco | | | | |
| PA Sat. | Admission | VASOACTIVE | Norepinephrine | Dopamine | Epinephrine | Vasopressin | Dobutamine | Milrinon |
| | Glucose | AGENTS: | | | | | | |
| | | (DOSE)- | | | | | | |
| | | (DOSE): | | | | | | l |

| ı | | RATORY VALUE | | | • | • | - | |
|---|---|---|---|---|---|---|---|---|
| HR | SBP | DBP | MAP | | | | | |
| RA/CVP | RV | PA | PCWP | CO Fick TD CCO | CI | СРО | PAPI | LVEDP |
| PA Sat. | VASOACTIVE<br>AGENTS:<br>(DOSE): | Norepinephrine | Dopamine | Epinephrine | Vasopressin | Dobutamine | Milrinone | Other: |

National CSI – Case Report Form – (v2.0) – July, 2018

| HR | SBP | ORATORY VALU | MAP | Troponin | Cr | AST | Hgb | Lactate |
|---|---|---|---|---|---|---|---|---|
| | 301 | | mai | Пороли | | | | Lucture |
| RA/CVP | RV | PA | PCWP | CO Fick TD CCO | СІ | СРО | PAPI | LVEDP |
| PA Sat. | VASOACTIVE<br>AGENTS: | Norepinephrine | Dopamine | Epinephrine | Vasopressin | Dobutamine | Milrinone | Other: |
| | (DOSE): | | | | | | | |
| | l | | | | | | | |
| HEMOD | NAMIC & LAB | ORATORY VALU | JES: 24 hou | rs Post-Impel | la Implant (C | ONLY if Impe | lla is runni | ng) |
| HR | SBP | DBP | MAP | Troponin | Cr | AST | Hgb | Lactate |
| RA/CVP | RV | PA | PCWP | со | СІ | СРО | PAPI | LVEDP |
| | | | | □ Fick □ TD<br>□ CCO | | | | |
| PA Sat. | VASOACTIVE<br>AGENTS: | Norepinephrine | Dopamine | Epinephrine | Vasopressin | Dobutamine | Milrinone | Other: |
| | (DOSE): | | | | | | | |
| Tin | ne & Date of In | AL FOLLOW UP npella Explant: MODYNAMIC SU reaned accordin | Time:<br>IPPORT:<br>g to: PA S | Sat □ Echo [<br>er: | | | | _ |
| Tin | ne & Date of In | npella Explant:<br>MODYNAMIC SU<br>reaned accordin | Time:<br>IPPORT:<br>g to: PA S | Sat □ Echo [ | | | | - |
| Tin<br>Wi | ne & Date of In<br>ANING OF HE!<br>Support was w | npella Explant:<br>MODYNAMIC SU<br>reaned accordin | Time:<br>IPPORT:<br>g to: | Sat □ Echo [<br>er: | □ RHC Hemo | dynamics | | - |

| Was the patient transferred to VAD/Transplant Center | Yes | No | N/A |
|---|---|---|---|
| If "Yes", DID THE PATIENT SURVIVE TO TRANSFER? | Yes | No | N/A |
| Did the patient have any additional support devices implanted post-index procedure? If "Yes", which device was used: | Yes | No | N/A |
| DID THE PATIENT SURVIVE TO DISCHARGE? | Yes | No | N/A |
| Was the patient discharged to hospice? | Yes | No | N/A |
| Did the patient experience any significant Impella-related NO Vascular Complications Hemolysis OTHER – Please explain: | | | |
| Did the patient require any blood transfusions? | ☐ Yes – # of | transfusions: | |
| Was any external form of vascular bypass performed to p | orovide lowe | | erfusion |
| during Impella (i.e. antegrade access, "up and over" perf | | | |
| during Impella (i.e. antegrade access, "up and over" perf | | | |
| during Impella (i.e. antegrade access, "up and over" perf | | | |
| during Impella (i.e. antegrade access, "up and over" perf No Yes – Please Explain: Please provide a brief description of the patient's hospita | al course (in | cluding signific | ant |
| during Impella (i.e. antegrade access, "up and over" perf No Yes – Please Explain: Please provide a brief description of the patient's hospita complications and discharge circumstances): | al course (in | cluding signific | ant |
| during Impella (i.e. antegrade access, "up and over" perf No Yes – Please Explain: Please provide a brief description of the patient's hospita complications and discharge circumstances): Please Explain: If the patient did not survive, please indicate the major of brain injury, worsening cardiogenic shock, patient/family | al course (in | cluding signific | ant |
| during Impella (i.e. antegrade access, "up and over" perf No Yes – Please Explain: Please provide a brief description of the patient's hospita complications and discharge circumstances): Please Explain: If the patient did not survive, please indicate the major of brain injury, worsening cardiogenic shock, patient/family | al course (in<br>ause of dear<br>wishes?) | cluding signific | ant<br>ing, anoxic |

# **Patient Exclusion Form**

# National Cardiogenic Shock Initiative

| | | | PATI | ENT EXCLU<br>(Version | JSION FORM<br>2.0) | |
|---|---|---|---|---|---|---|
| | Ple | ase con | | | CURE] email to: Nation or conce | |
| Hospit | al: | | | | | |
| Hospit | al - Cit | y, State | 2: | | | |
| Physici | ian: | | | | | |
| Date: | | | | | _ | |
| Age: _ | | | | | | |
| Gender | r: 🗆 N | /lale | ☐ Female | ☐ Other | | |
| Race: | □v | Vhite | □ Black | Hispanic | Other | |
| | | CARD | IOGENIC SHOC | K: Defined by th | ne presence of at lea | nce of STEMI or NSTEMI |
| | | va<br>□ Ev<br>el· | sopressors to r<br>ridence of end of<br>evated lactate | maintain SBP <u>&gt;</u> !<br>organ hypoperf<br>levels) | 90<br>usion (cool extremit | seline, or use of inotropes or<br>ties, oliguria or anuria, or<br>m2 or a cardiac power output |
| | | Patier | nt is supported | with Impella | | |
| | | Patier | nt undergoes P( | CI | | |
| National C | CSI — Patio | ent Exclusio | on Form — v2.0 — July, 2 | 1018 1 | | Continued on next page |

| | | CRITERIA: |
|---|---|---|
| YES | NO | |
| | | Evidence of Anoxic Brain Injury |
| | | Unwitnessed out of hospital cardiac arrest or any cardiac arrest in which ROSC is n |
| | | achieved in 30 minutes |
| | | IABP placed prior to Impella |
| | | Septic, anaphylactic, hemorrhagic, and neurologic causes of shock |
| | | Non-ischemic causes of shock/hypotension (pulmonary embolism, pneumothorax, |
| | | myocarditis, tamponade, etc.) |
| | | Active Bleeding |
| | | Recent major surgery |
| | | Mechanical Complications of AMI |
| | | Known left ventricular thrombus |
| | | Patient who did not receive revascularization |
| | | Mechanical aortic valve |
| | | Patient refused to sign consent for 1M & 1Y follow-up |
| Notes | 5: | |
| Comp | leted by | r: |
| SIGNA | TURE | |
| NAME | (PRINT | ED) |
| DATE | | |

# 30 Day Follow-Up Form

# National Cardiogenic Shock Initiative 30 Day Follow-Up

| | (Version 1.0) |
|---|---|
| | email this form via [SECURE] email to: <a href="MationalCSI@hfhs.org">NationalCSI@hfhs.org</a> , ail/call if there are any questions or concerns. |
| NCSI #: | |
| Hospital: | |
| Hospital - City, State: | |
| Date of Impella Implant: | <del></del> |
| Date of Follow-Up: | <del></del> |
| Patient Follow-Up — ≥ 30 Days | s from Date of Impella Implant: |
| Did the patient survive to 30 Days | s? |
| ☐ YES | |
| □ NO | |
| Unknown | |
| ☐ Patient Unavailable | |
| ☐ Refused | |
| Other: | |
| Point of Contact for Follow-up: | |
| ☐ Patient ☐ Spo | ouse 🗆 LAR/Proxy 🗆 Other: |
| Method of Follow-up: | |
| ☐ Phone Call | |
| ☐ Electronic Medical Rec | cord Review (patient signed-in for visit with ID at 30 or more days) |
| ☐ Mail | |
| ☐ Email | |
| Other: | |
| NOTES: | |
| Follow-up performed by: | |
| | Date: |
| National CSI – 30-Day Follow-Up—v1.0 – July, i | , 2018 |

# APPENDIX 6 1 Year Follow-Up Form

# National Cardiogenic Shock Initiative 1 Year Follow-Up

| | (Version 1.0) |
|---|---|
| Unon completion, pleas | se email this form via [SECURE] email to: NationalCSI@hfhs.org. |
| | email/call if there are any questions or concerns. |
| | and we will be any questions of concerns. |
| NCSI #: | |
| Hospital: | |
| Hospital - City, State: | |
| Date of Impella Implant: | |
| Date of Follow-Up: | |
| Patient Follow-Up; ≥ 365 D | ays from Date of Impella Implant: |
| Did the patient survive to 1-ye | <u> </u> |
| ☐ YES | |
| □NO | |
| Unknown | |
| ☐ Patient Unavailable | • |
| ☐ Refused | |
| ☐ Other: | |
| Point of Contact for Follow-up | p: |
| ☐ Patient ☐ Spouse [ | □ LAR/Proxy □ Other: |
| Method of Follow-up: | |
| ☐ Phone Call | |
| ☐ Electronic Medical | Record Review (patient signed-in for visit with ID at 365 or more days) |
| ☐ Mail | |
| ☐ Email | |
| ☐ Other: | |
| NOTES: | |
| | <del>_</del> |
| Signature: | Date: |